CLINICAL TRIAL: NCT01214590
Title: Preliminary Assessment of the Efficacy of the VascuActive™ Device on Diabetic Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VascuActive LTD (Industry)
Responsible Party: Yuval Avni, CEO, VascuActive
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAS-02
Record Dates: First submitted 2010-10-03; First posted 2010-10-05 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VascuActive Treatment (Experimental)
  Interventions: Device: VascuActive device

INTERVENTIONS:
Device: VascuActive device — self treatment by the patient, for 4 weeks, 3 sessions per day, approximately 30 minutes per session

SUMMARY:
The purpose of this study is to assess the safety and the preliminary efficacy of treatment by the VascuActive device on peripheral diabetic neuropathy, and to correlate this effect with physiologic changes.

Patients will undergo a 4-week period of home treatment by the VascuActive device, and will be monitored during this period and during a two-month follow-up period for the efficacy of the device in reducing neuropathic pain, sensation impairment and other signs and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus (type 1 or 2)
* Age 18 years or older
* No changes within the last 3 months in diabetes medications, pain management medications, and symptoms associated with diabetes
* Painful diabetic neuropathy > 3 months, but not more than 5 years
* Pain level ≥ 4 on an 11 point Numerical Pain Rating Scale in both feet (average of two measurements, at least 1 week apart, during the 2 weeks prior to first treatment)
* Loss of protective sensation by the 5.07 Semmes-Weinstein Monofilament (SWM, 10gr.) monofilament test (in both feet, at least at 3 out of 10 points in each foot)

Exclusion Criteria:

* Known or suspected radiculopathy (based on patient's record and anamnesis)
* Any painful condition that is difficult to distinguish from painful diabetic peripheral neuropathy
* Women at the age of fertility, who are pregnant, or plan pregnancy, or do not use contraceptive
* Severe cardiac disease or surgery within last 3 months, e.g., Acute Myocardial Infarction, Congestive Heart Failure grade 3 or higher
* Any major infectious, malignant or other severe systemic disease, including but not limited to Acquired Immune Deficiency Syndrome (AIDS), hepatitis, Creutzfeldt-Jakob disease
* Patient is incompetent to comply with study requirements (in the investigator's opinion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Diabetic neuropathic pain | 2, 4, 5, 12 weeks from start of treatment
  Pain will be assessed by several tools, including 11-point numeric scale, Brief Pain Inventory questionnaire, Pain relief scales (visual analog, categorical)

SECONDARY OUTCOMES:
Sensation impairment | 2, 4, 5, 12 weeks from start of treatment
  Touch sensation will be examined by the 5.07 Semmes-Weinstein monofilament (10 grams).
  Vibraion sensation will be examined by a 128Hz fork.
Nerve conduction velocity | 4, 12 weeks from start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Arie Bass, Prof., Principal Investigator — Assaf-Harofeh Medical Center; Robert Slater, Dr., Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Diabetic Foot Clinic, Tzrifin, Israel